CLINICAL TRIAL: NCT02264821
Title: Is Continuous Wound Infusion With Ropivacaine Better Than Intrathecal Morphine for Post-caesarean Analgesia? A Prospective, Randomized, Controlled, Double Blinded Study
Brief Title: Wound Infusion vs Spinal Morphine for Post-caesarean Analgesia
Acronym: Apcisaal
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr Madeleine Wilwerth (Other)
Responsible Party: Sponsor-Investigator, Dr Madeleine Wilwerth, Primary Investigator, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Apcisaal 01
Record Dates: First submitted 2014-08-25; First posted 2014-10-15 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-05

CONDITIONS: Post Caesarean Analgesia
Keywords: analgesia; caesarean; wound infiltration; intrathecal morphine.
MeSH Terms: conditions — Agnosia | interventions — Ropivacaine; Anesthetics, Local; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ropivacaine infiltration (Experimental): ropivacaine 2 mg/ml bolus 15 ml continuous 10 ml/h wound infusion and intrathecal saline
  Interventions: Drug: ropivacaine infiltration
- rachi morphine (Experimental): 100 µg intrathecal morphine and saline infiltration
  Interventions: Drug: intrathecal morphine
- placebo (Placebo Comparator): intrathecal saline and saline infiltration
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ropivacaine infiltration — wound infiltration
  Other Names: Naropin; local anesthetic
  Arms: ropivacaine infiltration
Drug: intrathecal morphine — 100 µg added to the spinal anaesthesia
  Other Names: spinal morphine
  Arms: rachi morphine
Drug: placebo — placebo in spinal anaesthesia and in wound infiltration
  Other Names: Nacl 0,9 %, saline solution
  Arms: placebo

SUMMARY:
The aim of this study is to compare effective analgesia with continuous wound infiltration of ropivacaine through multi-holed catheter or with morphine 100 mcg added intrathecally to spinal anesthesia, after elective Caesarean delivery.

DETAILED DESCRIPTION:
Double blind, 3 groups

* Control group: Rachi 0,1 ml saline, Infusion 300ml saline
* Group rachi-morphine: 0,1ml =100µg morphine/300ml saline
* Group KT: 0,1 ml saline/300 ml naropin 0.2%

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and more, ASA 1 or ASA 2, pregnant with at least 34 weeks of gestational age, admitted for a planned caesarian with a Pfannenstiel incision and having signed the informed consent form.

Exclusion Criteria:

* Refusal of the patient or contra-indication to locoregional anesthesia
* Allergy to the products used
* ASA 3
* ASA 4
* Sleep apnea syndrome and/or obesity (BMI > 35)
* Size inferior to 155cm
* existence of a language barrier

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2012-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Van der Linden, PhD, MD, Study Director — CHU Brugmann
Locations (1):
- Centre Hospitalier Universitaire Brugmann, Brussels, Belgium

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ropivacaine Infiltration | Rachi Morphine | Placebo
Started | 64 (Double Blind) | 64 (Double Blind) | 64 (Double Blind)
Completed | 63 | 61 | 58
Not Completed | 1 | 3 | 6
Not completed — Protocol Violation | 1 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine Infiltration | Rachi Morphine | Placebo | Total
Number analyzed (Participants) | 63 | 61 | 58 | 182
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [27 to 34] | 32 [28 to 34] | 32 [28 to 37] | 32 [27 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 61 | 58 | 182
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 63 | 61 | 58 | 182

OUTCOME MEASURES:

1. Primary Outcome: Duration of Effective Analgesia
Description: T0 until first request of morphine PCAIV
Time Frame: 30 hours after spinal injection T0
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Ropivacaine Infiltration | Rachi Morphine | Placebo
Number analyzed (Participants) | 63 | 61 | 58
minutes | 351 [227 to 594] | 380 [215 to 1527] | 247 [182 to 338]

2. Secondary Outcome: Incidence of Morphine Side Effects: Nausea, Vomiting, Pruritus.
Description: Is there a decrease of the incidence of morphine side effects such as nausea, vomiting, pruritus?
Time Frame: 30 hours after spinal injection
Reporting Status: Not Posted

3. Primary Outcome: Morphine Consumption
Description: Morphine consumption with PCAIV
Time Frame: 30 hours after spinal injection T0
Measure: Median (Inter-Quartile Range); unit: milligrammes
Arm/Group | Ropivacaine Infiltration | Rachi Morphine | Placebo
Number analyzed (Participants) | 63 | 61 | 58
milligrammes | 8 [4 to 20] | 4 [1 to 10] | 20.5 [9.5 to 31]

ADVERSE EVENTS:
Arm/Group | Ropivacaine Infiltration | Rachi Morphine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/61 | 0/58
Other Adverse Events (participants affected / at risk) | 61/63 | 61/61 | 58/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ropivacaine Infiltration (N=63) | Rachi Morphine (N=61) | Placebo (N=58)
Hypotension (Vascular disorders) | 22 | 23 | 30
Nausea and/or vomiting (Gastrointestinal disorders) | 10 | 18 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 31 | 35 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No